CLINICAL TRIAL: NCT04808323
Title: MRI-Guided Adaptive Radiation Therapy for Organ Preservation in Rectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William Hall, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00040139
Record Dates: First submitted 2021-02-16; First posted 2021-03-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Rectal Adenocarcinoma
Keywords: MR-guided radiation therapy; Rectal adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort A (Experimental): Radiation dose: 64 Gy over 32 fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to total dose of 64 Gy over 32 total fractions.
  Interventions: Drug: Capecitabine; Device: Initial Dose of Radiation before Dose Escalation; Device: Cohort A: Dose Escalation Radiation; Drug: FOLFOX
- Cohort B (Experimental): Radiation dose: 68 Gy over approximately 34 fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to 68 Gy over 34 total fractions.
  Interventions: Drug: Capecitabine; Device: Initial Dose of Radiation before Dose Escalation; Device: Cohort B: Dose Escalation Radiation; Drug: FOLFOX
- Cohort C (Experimental): Radiation dose: 72 Gy over 36 total fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to 72 Gy over 36 total fractions
  Interventions: Drug: Capecitabine; Device: Initial Dose of Radiation before Dose Escalation; Device: Cohort C: Dose Escalation Radiation; Drug: FOLFOX

INTERVENTIONS:
Drug: Capecitabine — 825 mg/m^2 twice daily during radiation therapy. (Fluorouracil (5-FU) may be used at the discretion of the treating medical oncologists.) This chemotherapy will be given during the initial radiation dose (50 Gy over 25 frac) and continue for Cohorts A, B, and C.
  Other Names: Xeloda
Device: Initial Dose of Radiation before Dose Escalation — 50 Gy over 25 frac.
Device: Cohort A: Dose Escalation Radiation — Cohort A will receive 14 Gy boost for a total of 64 Gy over 32 total fractions.
  Arms: Cohort A
Device: Cohort B: Dose Escalation Radiation — Cohort B will receive 18 Gy boost for a total of 68 Gy over 34 total fractions.
  Arms: Cohort B
Device: Cohort C: Dose Escalation Radiation — Cohort C will receive 22 Gy boost for a total of 72 Gy over 36 total fractions.
  Arms: Cohort C
Drug: FOLFOX — After the completion of radiation, subjects will receive up to eight cycles of systemic chemotherapy. (FOLFIRINOX may be used at the discretion of the treating medical oncologists.)
  Other Names: Oxaliplatin de Gramont; OxMdG

SUMMARY:
This study is a prospective, open-label, phase I design.

DETAILED DESCRIPTION:
Study Rationale: There are limited studies evaluating real-time adaptive radiation therapy for locally advanced (Stage I-III) rectal adenocarcinoma with the goal of accomplishing organ preservation. We are testing higher doses of radiation therapy, using a novel method of real-time adaptive MRI-based radiation therapy treatment.

Hypothesis: We hypothesize that adaptive magnetic resonance (MR) -guided radiation therapy will result in acceptable toxicity and that a maximum-tolerated dose can be determined in a phase I setting.

Intervention Description: The intervention in this circumstance is higher doses of radiation therapy focused within the tumor given using adaptive MR guidance. Radiation Doses being applied in this study:

Cohort A- 64 Gy over 32 fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to total dose of 64 Gy over 32 total fractions.

Cohort B- 68 Gy over approximately 34 fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to 68 Gy over 34 total fractions.

Cohort C- 72 Gy over 36 total fractions, prophylactic nodes treated to 50 Gy over 25 fractions, boost to tumor and radiologically positive nodes to 72 Gy over 36 total fractions.

Dose-Limiting Toxicity from Radiation Therapy: A dose-limiting toxicity (DLT) as per NCI CTCAE version 5. Specifically, this encompasses the need for additional treatments including the following: transfusion, invasive intervention, or hospitalization indicated. The presence of such a DLT would result in the halting of radiation therapy and impact on the dose levels of radiation therapy applied in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18.
2. Pathologically confirmed (histologic or cytological), adenocarcinoma of the rectum.
3. Determined on staging evaluation to be clinical stage I, II or III.
4. No concerning unequivocal or biopsy-proven metastatic disease. Patients are eligible with either no evidence of distant metastatic disease, or "equivocal" evidence of distant metastatic disease, as judged by the multidisciplinary tumor board. This "equivocal" definition can include small lung or liver lesions that are not able to be radiographically characterized otherwise.
5. Eastern Cooperative Oncology Group (ECOG) status 0-2 within 45 days of study entry.
6. History/physical examination, including collection of weight and vital signs within 45 days prior to start of treatment.
7. MR of the rectum is mandatory for staging and follow-up.
8. Chest CT scan within 45 days prior to study entry.
9. Radiation treatment planning abdominal CT. A mandatory pelvic MR will be done as a simulation (SIM) (ideally with interpretation). The CT SIM will not be done with interpretation. Ability to undergo abdominal MR scans for staging and radiation planning and follow-up is mandatory.
10. Laboratory values (CBC, Chem24) 45 days prior to treatment as follows:

    1. Carcinoembryonic antigen (CEA) (any value).
    2. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3.
    3. Platelets ≥50,000 cells/mm3.
    4. Hemoglobin ≥ 8.0 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
    5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 4 x upper limit of normal.
    6. Total bilirubin < 2 x upper normal mg/dL.
    7. Alkaline phosphatase < 4 x upper limit of normal.
11. Not on hemodialysis.
12. Ability to swallow oral medications.
13. Patients must be determined by medical oncology to be a candidate for systemic chemotherapy.
14. Patients must provide study-specific informed consent prior to study entry.
15. Negative serum pregnancy test (if applicable).
16. Women of childbearing potential and male participants who are sexually active must practice adequate contraception.

Exclusion Criteria:

1. Biopsy-proven distant metastatic disease or high clinical concern for metastatic disease and tumor conference consensus of stage IV disease.
2. Prior invasive malignancy (except nonmelanomatous skin cancer, noninvasive breast cancer (DCIS), or prostate cancer under active surveillance). Other malignancies are allowed if patient has been disease free for a minimum of three years
3. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
4. Any major surgery within 28 days prior to study entry, except colonic stent placement, intestinal diversion without resection or vascular access insertion.
5. Severe, active comorbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last six months.
   2. Transmural myocardial infarction within three months prior to study entry.
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
   4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
   5. Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function.
   6. Any unresolved intestinal obstruction.
   7. Acquired immune deficiency syndrome (AIDS), based upon current Centers for Disease Control and Prevention (CDC) definition. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because patients receiving antiretroviral therapy may experience possible pharmacokinetic interactions with required treatment medications, such as capecitabine.
   8. Absence of any significant medical comorbidity which would preclude the consideration of major intestinal surgery.
6. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during the course of the study and for women three months after study therapy is completed and for men six months after study therapy is completed. This exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
7. Participation in another interventional clinical treatment trial while on study (observational trials are permitted).
8. Patients taking nonprotocol-specified chemotherapy agents or immune-modulating agents for other medical conditions are not permitted to participate in this trial. Any medication questions should be reviewed by the PI.
9. Poor functional status such that patients are not able to be positioned for radiation treatments.
10. Gadolium allergy.
11. If age over 60, history of hypertension, diabetes or liver transplant, and glomerular filtration rate (GFR) at enrollment is < 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2029-01-20 (Estimated)

PRIMARY OUTCOMES:
The number of subjects in Cohort A with serious adverse events during radiation. | Up to 11.5-week period
  This will be measured by NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grades 3, 4 and 5 will be serious.
The number of subjects in Cohort B with serious adverse events during radiation. | Up to 11.5-week period
  This will be measured by NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grades 3, 4 and 5 will be serious.
The number of subjects in Cohort C with serious adverse events during radiation. | Up to a 12.1-week period.
  This will be measured by NCI Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grades 3, 4 and 5 will be serious.

SECONDARY OUTCOMES:
The number of subjects in Cohort A with a complete clinical response (CCR) to treatment. | 31.5 weeks
  Four weeks following completion of chemotherapy, radiation therapy (RT), and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  CCR is defined as meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis.
The number of subjects in Cohort B with a complete clinical response (CCR) to treatment. | 31.5 weeks
  Four weeks following completion of chemotherapy, RT, and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  CCR is defined as meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis.
The number of subjects in Cohort C with a complete clinical response (CCR) to treatment. | 32.1 weeks
  Four weeks following completion of chemotherapy, RT, and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  CCR is defined as meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis.
The number of subjects in Cohort A with a noncomplete response (NCR) to treatment. | 31.5 weeks
  Four weeks following completion of chemotherapy, RT, and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  A noncomplete clinical response is defined as any state not meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis. If the tumor site does not meet the above criteria, the patient will be classified as noncomplete response (NCR).
The number of subjects in Cohort B with a noncomplete response (NCR) to treatment. | 31.5 weeks
  Four weeks following completion of chemotherapy, RT, and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  A noncomplete clinical response is defined as any state not meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis. If the tumor site does not meet the above criteria, the patient will be classified as noncomplete response (NCR).
The number of subjects in Cohort C with a noncomplete response (NCR) to treatment. | 32.1 weeks
  Four weeks following completion of chemotherapy, RT, and neoadjuvant systemic chemotherapy, the patient will be evaluated by the study surgeon to assess local response.
  A noncomplete clinical response is defined as any state not meeting the following criteria:
  1. No palpable tumor on digital exam.
  2. Endoscopic evaluation consistent with the following.
     1. Flat scar with no ulceration and intact mucosa.
     2. Disappearance of neoplastic pit pattern without use of magnification.
     3. Disappearance of neoplastic nodule or stenosis. If the tumor site does not meet the above criteria, the patient will be classified as noncomplete response (NCR).
Circulating tumor deoxyribonucleic acid (ctDNA) | Baseline, 12.1 weeks, 32 weeks, one year and two years.
  Blood samples (10 mL each time) will be collected. ctDNA is measured in percentage: variant allele fraction percentage. For simplicity this will be reported at baseline, the end of radiation, the end of neoadjuvant treatment and annually for two years.
The number of subjects with dose-limiting toxicities in Cohort A. | 11.5-week period
  Number of subjects experiencing a dose-limiting toxicity (DLT) as per NCI CTCAE version 5, encompasses the need for additional treatments including the following: transfusion, invasive intervention, or hospitalization indicated. The presence of such a DLT would result in the halting of radiation therapy and impact on the dose levels of radiation therapy applied in the trial.
The number of subjects with dose-limiting toxicities in Cohort B. | 11.5-week period
  Number of subjects experiencing a dose-limiting toxicity (DLT) as per NCI CTCAE version 5, encompasses the need for additional treatments including the following: transfusion, invasive intervention, or hospitalization indicated. The presence of such a DLT would result in the halting of radiation therapy and impact on the dose levels of radiation therapy applied in the trial.
The number of subjects with dose-limiting toxicities in Cohort C. | 12.1- week period
  Number of subjects experiencing a dose-limiting toxicity (DLT) as per NCI CTCAE version 5, encompasses the need for additional treatments including the following: transfusion, invasive intervention, or hospitalization indicated. The presence of such a DLT would result in the halting of radiation therapy and impact on the dose levels of radiation therapy applied in the trial.
Change from baseline in the EQ-5D-SL quality of life questionnaire | Baseline and up to 12.1 weeks.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (coded as 1), slight problems (coded as 2), moderate problems (coded as 3), severe problems (coded as 4) and extreme problems (coded as 5). The score is expressed as a five-digit number. The second part of the instrument (EQ VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (score of 100) and 'The worst health you can imagine' (score of 0).
Change from baseline in the Memorial Sloan Kettering Bowel Function Index (MSKCC BFI) Score | Baseline and up to 12.1 weeks.
  The MSKCC BFI comprises 18 items covering the frequency of various symptoms and is divided into three sub-scales and four single items. It is scored on a 5-point Likert scale ranging from "always" to "never". The sub-scales scores are summarised as: A 6-item frequency sub-scale (6-30), a four-item dietary sub-scale (4-20), and a four-item urgency sub-scale (4-20). A global score can be calculated as the sum of the sub-scale scores. A total score (possible score range 18-90) can be calculated by adding all the item scores (sub-scale scores plus single item scores). A higher score indicates better bowel function.
Change from baseline in the Wexner Fecal Incontinence Score | Baseline and up to 12.1 weeks.
  This scoring system cross-tabulates frequencies and different anal incontinence presentations (Gas/Liquid/Solid/Pad use/Need for lifestyle alterations) and sums the returned score to a total of 0-20 (where 0 = perfect continence and 20 = complete incontinence). Each of the incontinence presentations is graded equally.

CONTACTS AND LOCATIONS:
Overall Officials: William Hall, MD, Principal Investigator — Medical College of Wisconsin; Carrie Peterson, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No